CLINICAL TRIAL: NCT01897376
Title: The Comparative Effectiveness of Pfannenstiel Versus Vertical Skin Incision in Preventing Wound Complications After Cesarean Delivery in Morbidly Obese Women: a Randomized Clinical Trial.
Brief Title: Cesarean Skin Incision Trial
Acronym: C-SIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: The University of Texas Medical Branch, Galveston (Other)
Responsible Party: Principal Investigator, Caroline Carter Marrs, MD, M.D., The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: C-SIT
Record Dates: First submitted 2013-07-08; First posted 2013-07-12 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2017-06

CONDITIONS: Wound Complication
Keywords: wound; infection; cesarean delivery; obesity
MeSH Terms: conditions — Wounds and Injuries; Infections; Obesity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Pfannenstiel incision (Other)
  Interventions: Procedure: Pfannenstiel incision
- vertical skin incision (Other)
  Interventions: Procedure: vertical skin incision

INTERVENTIONS:
Procedure: Pfannenstiel incision — Pfannenstiel incision at time of cesarean section
  Arms: Pfannenstiel incision
Procedure: vertical skin incision — vertical skin incision at time of cesarean section
  Arms: vertical skin incision

SUMMARY:
The purpose of this study is to determine if there is a difference between Pfannenstiel and midline vertical skin incision at time of cesarean section in preventing wound complications in the morbidly obese patient. This is a comparative effectiveness study of two commonly-used skin incisions. The investigators plan to enroll morbidly obese obstetrical patients upon admission and randomize them to one of the above incision types in the operating room. The investigators will follow them for 6 weeks post-op to evaluate for wound complications. There is minimal risk to the participant as both incision types are acceptable in current obstetrical practice. There is no direct benefit to the patient.

Currently, there is no level I evidence to support either Pfannenstiel or midline vertical skin incision in the prevention of wound complications in the obese patient undergoing cesarean section. Therefore, current practice is for the surgeon to make the decision based on preference and weighing theoretic risks. Therefore, there is clinical equipoise. Cesarean section is a very common procedure, with a national rate of 32% of all live births in 2007. Not only does obesity increase the expectant mother's risk of a cesarean section, it is also a well recognized risk factor for wound complication. The cesarean wound complication rate in the morbidly obese population at the University Of Texas at Houston - Memorial Hermann Hospital Texas Medical Center in 2011 was roughly twenty times as high as the normal weight population, 28% compared to 1.4%. Results from this study could be extrapolated in the future to affect lower post-operative morbidity, higher patient satisfaction, less antibiotic use, shorter hospital stay, and overall lower health care costs.

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant women undergoing cesarean delivery for any indication, regardless of number of prior cesarean deliveries
2. Age 18-50 years
3. BMI of 40 kg/m2 or more

Exclusion Criteria:

1. Underlying infection such as chorioamnionitis
2. Rupture of membranes over 18 hours prior to cesarean section ,

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 228 (Actual)
Dates: Start 2013-07; Primary Completion 2017-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
composite wound complication | 6 weeks post-op
  includes surgical site infection as defined by the Centers for Disease Control, as well as seromas, cellulitis, and wound separations

CONTACTS AND LOCATIONS:
Overall Officials: Caroline C Marrs, MD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (2):
- United States (2):
  - UTMB, Galveston, Texas
  - Memorial Hermann Hospital Texas Medical Center, Houston, Texas

REFERENCES:
- [Derived] Marrs C, Blackwell S, Hester A, Olson G, Saade GR, Faro J, Pedroza C, Sibai B. Pfannenstiel versus Vertical Skin Incision for Cesarean Delivery in Women with Class III Obesity: A Randomized Trial. Am J Perinatol. 2019 Jan;36(1):97-104. doi: 10.1055/s-0038-1667287. Epub 2018 Jul 30. PMID 30060292